CLINICAL TRIAL: NCT07406321
Title: Efficacy of Cognitive Bias Modification Itervention in Young Adult With Social Anxiety
Brief Title: Brief Interpretation Bias Modification for Social Anxiety Disorder in Pakistani Young Adults: An Experimental Evaluation
Acronym: BIBM-SAD-PYA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ather Mujitaba (Other)
Responsible Party: Sponsor-Investigator, Ather Mujitaba, PhD Scholar, University of Gujrat
Organization: University of Gujrat (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOG/ORIC/2025/342
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Social Anxiety Disorder; Interpretation Bias
Keywords: interpretation bias modification; Word-Sentence Association Paradigm; Social Anxiety Disorder; Pakistan Young Adult; Cogntive Bias Modification
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Parallel Assignment.
Who Masked: Participant
Masking Description: Participants are unaware of arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpretation Bias Modification (Experimental): Single-session Word-Sentence Association Paradigm training with performance-contingent feedback across 220 trials in two 110-trial blocks; each block includes 70 social ambiguity trials and 40 non-social fillers. Correct feedback follows benign endorsement or threat rejection; incorrect feedback follows threat endorsement or benign rejection.
  Interventions: Behavioral: WSAP-based interpretation bias modification
- Interpretation Control Condition (Active Comparator): Matched Word-Sentence Association Paradigm exposure with identical stimulus timing and response demands, feedback delivered on 50 percent of trials without contingency, favoring benign over threat interpretations.
  Interventions: Behavioral: WSAP interpretation control condition

INTERVENTIONS:
Behavioral: WSAP-based interpretation bias modification — Single-session Word-Sentence Association Paradigm training with performance-contingent feedback across 220 trials in two 110-trial blocks; each block includes 70 social ambiguity trials and 40 non-social fillers. Correct feedback follows benign endorsement or threat rejection; incorrect feedback follows threat endorsement or benign rejection.
  Arms: Interpretation Bias Modification
Behavioral: WSAP interpretation control condition — Matched Word-Sentence Association Paradigm exposure with identical stimulus timing and response demands, feedback delivered on 50 percent of trials without contingency favoring benign over threat interpretations.
  Arms: Interpretation Control Condition

SUMMARY:
This randomized, single-blind trial tests whether one session of interpretation bias modification reduces immediate social-evaluative anxiety and shifts interpretation bias in Pakistani university students aged 18 to 25 years with elevated social anxiety. Participants are assigned to either feedback-contingent interpretation bias modification or a structurally matched interpretation control condition. Primary and secondary outcomes are assessed before and after the intervention session using short-form state-trait anxiety measures and Word-Sentence Association Paradigm endorsement indices.

DETAILED DESCRIPTION:
Social anxiety in young adults is maintained in part by a tendency to interpret ambiguous social information as threatening. The study evaluates a behavioral interpretation training procedure delivered with OpenSesame, using trial-by-trial responses to ambiguous social sentences preceded by threat or benign prime words. In the experimental arm, feedback contingently reinforces benign endorsements and threat rejections. In the control arm, exposure and timing are matched but feedback is noncontingent and presented on half of trials. The design is a parallel two-arm randomized pretest-posttest trial with participant masking to assignment. Assessment includes the 5-item state and 5-item trait short-form State-Trait Anxiety Inventory totals and Word-Sentence Association Paradigm threat and benign endorsement proportions. The mechanistic hypothesis is that feedback-consistent learning increases benign interpretations and reduces threat interpretations, which is associated with lower post-session state anxiety. The trial was conducted as part of a PhD thesis at the University of Gujrat under formal institutional approvals.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 25 years
* Social Phobia Inventory score greater than 19
* at least moderate severity on the DSM-5-TR Severity Measure for Social Anxiety Disorder-Adult
* able to read study materials
* provides written informed consent.

Exclusion Criteria:

* clinically elevated depressive symptoms on Beck Depression Inventory-II at or above prespecified cutoff [above 16]
* clinically elevated general anxiety symptoms on the Beck Anxiety Inventory at or above prespecified cutoff [ above 20]
* current medical or psychiatric condition likely to interfere with safe or valid participation
* prior participation in this trial.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
short version of the Spielberger State-Trait Anxiety Inventory | Baseline (pre-intervention, same visit) and immediate post-intervention after the single-session training (same visit, approximately 30 to 60 minutes after intervention)
  The primary outcome is within-participant change in state anxiety measured with the 5-item short-form State-Trait Anxiety Inventory state subscale (STAIS-5). Items are summed to a total score, with higher scores indicating greater state anxiety. The primary comparison is the between-group difference in change score (IBM versus ICC).
Spielberger short-form State-Trait Anxiety Inventory (S-STAI) | Baseline pre-intervention and immediate post-intervention in the same visit (approximately 30 to 60 minutes after training starts).
  Difference between post-session and baseline STAIS-5 total score; higher scores indicate greater state anxiety.

SECONDARY OUTCOMES:
Change in Word-Sentence Association Paradigm threat endorsement rate. | Baseline pre-intervention and immediate post-intervention in the same visit.
  Proportion of threat word-sentence pairings endorsed as related; lower values indicate less threat-consistent interpretation. Used as interpretation bias metrices.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Riaz Riaz, PhD, Principal Investigator — University of Gujrat
Locations (1):
- University of Gujrat, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are not available at this stage because the trial is ongoing and data collection is not complete. After study completion, data cleaning, and primary reporting, the team will determine whether de-identified individual participant data can be shared in line with institutional approvals, participant consent, and applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Supporting documents will be considered for release after final study completion and primary thesis/manuscript reporting. The exact release start date and duration have not yet been finalized and will be updated in the registry record after completion.
Access Criteria: Access procedures are not yet finalized. Any future sharing will be limited to de-identified materials and will require a reasonable scientific request, ethical use, and institutional approval as applicable. Final criteria will be added after study completion.
URL: https://uog.edu.pk/faculty/jst57cea53bf24cd/saima-riaz

REFERENCES:
- [Result] 1. Hofmann SG. Cognitive factors that maintain social anxiety disorder: a comprehensive model and its treatment implications. Cogn Behav Ther. 2007;36(4):193-209. doi:10.1080/16506070701421313. 2. Ejaz B, Muazzam A, Anjum A, Pollock G, Nawaz R. Measuring the scale and scope of social anxiety among students in Pakistani higher education institutions: an alternative social anxiety scale. Sustainability. 2020;12(6):2164. doi:10.3390/su12062164. 3. Rapee RM, Heimberg RG. A cognitive-behavioral model of anxiety in social phobia. Behav Res Ther. 1997;35(8):741-756. doi:10.1016/S0005-7967(97)00022-3. 4. Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA. Manual for the State-Trait Anxiety Inventory (Form Y). Palo Alto (CA): Consulting Psychologists Press; 1983. 5. Beard C, Amir N. Negative interpretation bias mediates the effect of social anxiety on state anxiety. Cognit Ther Res. 2010;34(3):292-296. doi:10.1007/s10608-009-9258-6. 6. Hallion LS, Ruscio AM. A meta-analysis of the effect of cognitive bias modification on anxiety and depression. Psychol Bull. 2011;137(6):940-958. doi:10.1037/a0024355. 7. MacLeod C, Mathews A. Cognitive bias modification approaches to anxiety. Annu Rev Clin Psychol. 2012;8:189-217. doi:10.1146/annurev-clinpsy-032511-143052. 8. Amir N, Bomyea J, Beard C. The effect of a single-session interpretation modification on attention bias in socially anxious individuals. J Anxiety Disord. 2010;24(2):178-182. doi:10.1016/j.janxdis.2009.10.005. 9. Beard C, Amir N. Interpretation in social anxiety: when meaning precedes ambiguity. Cognit Ther Res. 2009;33(4):406-415. doi:10.1007/s10608-009-9235-0. 10. Gonsalves M, Whittles RL, Weisberg RB, Beard C. A systematic review of the word sentence association paradigm (WSAP). J Behav Ther Exp Psychiatry. 2019;64:133-148. doi:10.1016/j.jbtep.2019.04.003. 11. Connor KM, Davidson JRT, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). Br J Psychiatry. 200